CLINICAL TRIAL: NCT03413579
Title: Multicenter Randomised Double-blind Study to Compare HR3 or Placebo in Combination With Cisplatin-navelbine for Patients With Cervical Carcinoma, Followed in Case of Progression by a Second Line.
Brief Title: Evaluate Efficacy of the Association Nimotuzumab(HR3) /Cisplatin-Vinorelbine on Patients With Cervical Carcinom
Acronym: CIMAHOPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: El Kendi Pharmaceuticals Manufacturing Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIMA-I3-05D143-01
Record Dates: First submitted 2018-01-11; First posted 2018-01-29 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2020-03

CONDITIONS: Cervical Cancer
Keywords: Cervix; Oncology,; hR3,; Nimotuzumab,; Chemotherapy,; Survival; Monoclonal antibody; RECIST; Cisplatin; Vinorelbine; Paclitaxel; Carboplatine; Randomisation; Placebo; cancer; cimahope
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms | interventions — nimotuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nimotuzumab (Experimental): Injection of 200 mg of Nimotuzumab (weekly during 18 weeks), in combination with chemotherapy (6 cycles, every 21 days: 70 mg / m2 Cisplatin and Vinorelbine 60 mg / m2 (Per Os) at day 1 and day 8.
  The objective of the present study is to assess the overall survival of patients after administration of Nimotuzumab hR3 monoclonal antibodies (combined with a chemotherapy) in the treatment of patients with cervix epithelial tumors as first-line treatment.
  After the first line , a 200mg dose of hR3 monoclonal antibodies will be given every 14 days until progress.
  A second -line chemotherapy is proposed, this is based on Carboplatin (CBP) at AUC of 6, and Paclitaxel (Txl) 175 mg / m2 / SC as 3 hour infusion, every 3 weeks, concomitant with the administration of hR3, every 14 days, until a toxicity limit or an ECOG status greater than 3 appears.
  Interventions: Biological: Nimotuzumab ( h-R3)
- Placebo (Placebo Comparator): Injection of the Placebo in the same procedures (weekly during 18 weeks), in combination with chemotherapy (6 cycles, every 21 days: 70 mg / m2 Cisplatin and Vinorelbine 60 mg / m2 (Per Os) at day 1 and day 8.
  After the first line , a 200mg dose of hR3 monoclonal antibodies will be given every 14 days until progress.
  A second -line chemotherapy is proposed, this is based on Carboplatin (CBP) at AUC of 6, and Paclitaxel (Txl) 175 mg / m2 / SC as 3 hour infusion, every 3 weeks, concomitant with the administration of hR3, every 14 days, until a toxicity limit or an ECOG status greater than 3 appears.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Nimotuzumab ( h-R3) — Humanized monoclonal antibody
  Other Names: CIMAHOPE
  Arms: Nimotuzumab
Other: Placebo
  Arms: Placebo

SUMMARY:
The objective of the present study is to estimate the overall survival of patients with cervical cancer after the administration of monoclonal antibody (mAb) Nimotuzumab (hR3) in combination with chemotherapy of first intention. Patients will be randomized in two parallel treatment groups. The first group will receive a dose of 200 mg of monoclonal antibody anti-hR3 (weekly during 18 weeks), combined with a chemotherapy (6 cycles, every 21 days of Cisplatin 70mg/m2, Vinorelbine 60 mg/m2 (Per Os) at D1 and D8 and then 80mg / m2. The second group will receive a placebo in combination with the same chemotherapy regimen as the first group.

At the end of the first intention chemotherapy treatment, a dose of maintenance of Nimotuzumab will be administered at the dose of 200mg every 14 days until progression. A second chemotherapy in the second intention is proposed, this one is based on Carboplatin ( CBP) in an AUC (area under curve) of 6, and Paclitaxel (Txl) in 175 mg / m2 / BSA (body surface area ) in drip of 3 hours, every 3 weeks, concomitant with the administration of hR3, every 14 days, until a limit of toxicity or an ECOG (Eastern Cooperative Oncology Group) status superior to 3, appears.

DETAILED DESCRIPTION:
The objective of the present study is to assess the overall survival of patients after administration of Nimotuzumab hR3 monoclonal antibodies (combined with a chemotherapy) in the treatment of patients with cervix epithelial tumors as first-line treatment.

The patients included will be divided into two treatment groups. The first group receive a 200 mg dose of hR3 monoclonal antibody (weekly for 18 weeks), and chemotherapy (6 cycles, every 21 days: Cisplatin (CDDP) 70 mg / m2 on day 1, Vinorelbine 60 mg / m2 on day 1 and day 8) and then 80mg / m2. The second group receive a placebo in addition to the listed chemotherapy.

After the first line , a 200mg dose of hR3 monoclonal antibodies will be given every 14 days until progress.

A second -line chemotherapy is proposed, this is based on Carboplatin (CBP) at AUC of 6, and Paclitaxel (Txl) 175 mg / m2 / SC as 3 hour infusion, every 3 weeks, concomitant with the administration of hR3, every 14 days, until a toxicity limit or an ECOG status greater than 3 appears.

The survival overall will be considered as the main variable of the response and survival without progression from the antitumor response, the toxicity assessment and the quality of life will be the secondary variables. In addition, the effects may arise during treatment will be identified, and tumor biopsy markers such as, EGF-R and HPV will be determined and those of p53, Ki67 and Bcl-2 by immunohistochemistry (IHC).

It is expected to achieve a difference in survival between the treatment groups of 6.5 vs 10.5 months (0.278 vs 0.62) in favor of the group with mAb hR3.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 to 75, including both limits.
* Patients who give their written consent to participate to the study.
* Chemonaive patients with local cervical cancer and / or persistent or recurrent metastatic disease with measurable disease (RECIST criteria) by a physical examination (scanner or MRI).

A confirmation by biopsy is necessary in case there is a single lesion less than 2 cm.

* Patients who had pelvic CT + radiotherapy may also be included in the study (concomitant chemotherapy as a radiotherapy stabilizer).
* Patients having a histopathological report: epidermoid carcinoma, adenocarcinoma, adenosquamous carcinoma and / or clear cells carcinoma.
* Patients with an ECOG score between 0-2
* Patients with a life expectancy greater than six months.
* Patients with Left Ventricular Ejection Fraction (LVEF) ≥50%, through Echocardiography.
* Patients with normal function of organs and bone marrow, defined by the following parameters:

  * Haemoglobin ≥ 9 g / dL
  * White Blood cell ≥ 4000 /mm3
  * Absolute neutrophil count≥ 1500 /mm3
  * Platelet count≥ 100000 /mm3
  * Total bilirubin up to 1.5 the upper limit of normal (ULN)
  * Albumin ≥ 2 g/dL (3,5 - 5,0 g /dl)
  * Serum Glutamopyruvate Transférase (SGPT) and SErum Glutamooxaloacetate Transferase (SGTO) < or = 2.5 ULN
  * Serum creatinine within the normal limits and the calculation of glomerular filtration according to Cockcroft formula ≥ 60ml and according to MDRD formula for patients whose age is 70 years ≥ 60ml . Glomerular filtration will be performed only on clinical discretion for patients suspected to have a kidney problem. (The normal laboratory values will be appropriate to the techniques and equipment used in the place where they are done).
* The determination or expression of EGF-R (epidermal growth factor receptor), p53, Ki67 and Bcl-2 by immuno-histochemistry in the primary tumor before treatment integrated in a paraffin block.

The results are not an inclusion criterion, but will be evaluated as an indicator of prognostic response in the final assessment.

Exclusion Criteria:

* Pregnant or breastfeeding patients
* Patients with small cells and / or neuroendocrine cervical cancer.
* Patients receiving another onco-specific drug, for other clinical trial,
* Patients with a history of allergy attributed to chemical or biological compounds similar to the monoclonal antibody being evaluated or to chemotherapeutic agents.
* Patients having uncontrolled intercurrent diseases, including active infections, symptomatic congestive heart failure , unstable angina, cardiac arrhythmia, decompensated diabetes, uncontrolled hypertension and psychiatric disorders.
* Patients having a second tumor . Excepting for those receiving appropriate therapy for skin cancer (basal or squamous)
* Previous or concomitant malignancy with exception for non-melanoma skin carcinomas
* Patients having special conditions or circumstances that could significantly limit the complete follow up of the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 37 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Overall survival in patients who received hR3 mAb treatment combined with Chemotherapy | Calculated from patient randomisation to death (36 months)

SECONDARY OUTCOMES:
Antitumor Response | up to 24months (every 3 months)
Duration of response | from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
Time to progression | Time from randomization until objective tumor progression assessed up to 60 months
Progression-free survival | Time from randomization until disease progression or death, assessed up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed MECHETI, MD., Study Director — El Kendi, Part of MS Pharma, Manufacturing Company
Locations (5):
- Algeria (5):
  - Centre Pierre et Marie Curie (CPMC), Algiers
  - CAC Annaba, Annaba
  - CAC Batna, Batna City
  - CHU Frantz Fanon, Blida
  - CHU Sidi Belloua, Tizi Ouzou